CLINICAL TRIAL: NCT06860633
Title: Treatment of Myasthenia Gravis Exacerbation or Crisis With Efgartigimod: A Single Arm, Open Label Prospective Cohort Study
Brief Title: Treatment of Myasthenia Gravis Exacerbation or Crisis With Efgartigimod
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-0158
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Myasthenia Gravis Crisis; Myasthenia Gravis Exacerbations; AChR Myasthenia Gravis
Keywords: myasthenia exacerbation; efgartigimod
MeSH Terms: interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Efgartigimod (Experimental): Participants receive 4 doses of efgartigimod via intravenous (IV) infusion over the course of the study on days 1, 4, 11 and 18.
  Interventions: Drug: Efgartigimod

INTERVENTIONS:
Drug: Efgartigimod — Dose of 10 mg/kg for IV infusion on days 1, 4, 11 and 18
  Other Names: Vyvgart

SUMMARY:
This study plans to learn more about if the drug efgartigimod can be used in the hospital to treat exacerbations in participants with myasthenia gravis (MG). Efgartigimod has been approved by the FDA for ongoing (chronic) treatment of generalized MG in adult patients who are anti-acetylcholine receptor (AChR) antibody positive but has not been studied in the treatment of worsening weakness requiring hospital admission (known as "exacerbation"). This investigation aims to see if using efgartigimod in this way improves symptoms and recovery from exacerbation, and how it affects certain MG markers in the blood. The main questions it aims to answer are:

* Is efgartigimod effective as a hospital-administered acute therapy for participants with worsening MG (MG exacerbation) who require hospitalization?
* Will efgartigimod lead to clinical improvement with a similar reduction in validated research scales, such as the Quantitative MG (QMG) scale, as standard of care therapies?

Participants will receive 4 doses of efgartigimod over the course of 4 weeks with an additional follow-up visit at the clinic.

DETAILED DESCRIPTION:
Efgartigimod is thought to work by reducing circulating IgG antibodies, including the antibodies that cause MG. One of the currently used treatments for MG exacerbation, called plasma exchange (PLEX), is also thought to work by reducing antibody levels by filtering blood through a machine similar to those used in dialysis for kidney failure. Because of the similarities between how these two treatments work, there is reason to believe that efgartigimod may also be helpful in treating MG exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ age 18 years with known generalized MG as identified by characteristic signs of generalized MG on clinical assessment and positive serology for AchR antibodies as well as one of the following:

  1. Documented positive response to cholinesterase inhibitors such as pyridostigmine or edrophonium
  2. Abnormal decrement on slow repetitive nerve stimulation testing
  3. Abnormal single fiber EMG
* Evidence of worsening weakness requiring hospital admission for stabilization and change in therapy as determined by a neuromuscular expert including:

  1. Quantitative Myasthenia Gravis (QMG) scale ≥ 11
  2. MG-ADL score ≥ 6
  3. Worsening weakness that is unlikely to be ameliorated by adjustment of current medications including impaired respiratory status, dysarthria, dysphagia, difficulty chewing, limb weakness, diplopia, ptosis.
* Ability to sign consent and be enrolled within 24 hours of hospital admission. For participants transferred to University of Colorado Hospital, the time of admission/presentation to the outside hospital is counted towards this 24-hour cap.

Exclusion Criteria:

* MG worsening thought to be related to active infection or due to medications (e.g. fluoroquinolone or aminoglycoside antibiotics, magnesium, chloroquine derivatives)
* Intubation prior to ability to sign informed consent or intubation within 24 hours of hospitalization
* Use of IVIG within 2 weeks, or having undergone plasma exchange or received efgartigimod in the 4 weeks prior to admission
* Current ongoing use of ravulizumab or eculizumab (monoclonal antibody C5-complement inhibitors).
* Other medical conditions that, in the opinion of the investigator and treating clinicians, might interfere with the validity of assessment measures used in the study (e.g. steroid myopathy, CNS pathology, severe arthritis, fractures, etc.). This criterion is a standard exclusion in MG trials and relates solely to other conditions that reduce muscle power or range of motion and would thus worsen scores on assessment measures like the QMG due to non-MG conditions.
* Known history of coagulopathy, blood clotting, recent severe bleeding (e.g. GI bleed).
* Pregnancy or breastfeeding. Pregnancy must be excluded for all potential participants who are able to become pregnant prior to initiation of treatment.
* IgG levels < 600mg/dL
* Evidence of active or chronic Hepatitis B infection, untreated Hepatitis C infection, HIV with low CD4 (<200) count.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Quantitative Myasthenia Gravis (QMG) score at day 11 | Baseline, Day 11
  The Quantitative Myasthenia Gravis (QMG) is a scoring system that quantifies disease severity by measuring ocular, bulbar, respiratory and limb strength. The total scores range from 0 to 39, with higher scores indicating greater disease severity.

SECONDARY OUTCOMES:
Percentage of participants requiring rescue therapy with Plasma Exchange (PLEX) or Intravenous Immunoglobulin (IVIG) | During hospitalization, approximately 7 days
  Number of participants requiring rescue therapy with Plasma Exchange (PLEX) or Intravenous Immunoglobulin (IVIG) over number of total participants
Change from baseline in Myasthenia Gravis Activities of Daily Life (MG-ADL) scale at day 18 | Baseline, Day 18
  The Myasthenia Gravis Activities of Daily Life (MG-ADL) is a questionnaire administered verbally that measures MG symptoms and functional activities related to activities of daily living. The summative total scores range from 0 to 24, with higher scores indicating greater disease severity.
Change from baseline in Myasthenia Gravis Activities of Daily Life (MG-ADL) scale at day 32 | Baseline, Day 32
  The Myasthenia Gravis Activities of Daily Life (MG-ADL) is a questionnaire administered verbally that measures MG symptoms and functional activities related to activities of daily living. The summative total scores range from 0 to 24, with higher scores indicating greater disease severity.
Change from baseline in Myasthenia Gravis Manual Muscle Test (MG-MMT) at day 11 | Baseline, Day 11
  The Myasthenia Gravis Manual Muscle Test (MG-MMT) is an assessment that assigns numerical values to the presence of mild, moderate or severe weakness for specific muscle groups that may be affected by MG. The summative total scores range from 0 to 120, with higher scores indicating greater disease severity.
Change from baseline in Myasthenia Gravis Manual Muscle Test (MG-MMT) at day 18 | Baseline, Day 18
  The Myasthenia Gravis Manual Muscle Test (MG-MMT) is an assessment that assigns numerical values to the presence of mild, moderate or severe weakness for specific muscle groups that may be affected by MG. The summative total scores range from 0 to 120, with higher scores indicating greater disease severity.
Change from baseline in Myasthenia Gravis Manual Muscle Test (MG-MMT) at day 32 | Baseline, Day 32
  The Myasthenia Gravis Manual Muscle Test (MG-MMT) is an assessment that assigns numerical values to the presence of mild, moderate or severe weakness for specific muscle groups that may be affected by MG. The summative total scores range from 0 to 120, with higher scores indicating greater disease severity.
Change from baseline in Myasthenia Gravis Quality of Life-15 Revised (MG-QOL15r) at day 18 | Baseline, Day 18
  The Myasthenia Gravis Quality of Life-15 Revised (MG-QOL15r) is a scale that measures perceived limitations to fifteen different activities due to MG. Individual items are score 0 (not at all) to 4 (quite a bit). The summative total scores range from 0 to 60, with higher scores representing worse quality of life.
Change from baseline in Myasthenia Gravis Quality of Life-15 Revised (MG-QOL15r) at day 32 | Baseline, Day 32
  The Myasthenia Gravis Quality of Life-15 Revised (MG-QOL15r) is a scale that measures perceived limitations to fifteen different activities due to MG. Individual items are score 0 (not at all) to 4 (quite a bit). The summative total scores range from 0 to 60, with higher scores representing worse quality of life.
Change from baseline in the Quantitative Myasthenia Gravis (QMG) score at day 4 | Baseline, Day 4
  The Quantitative Myasthenia Gravis (QMG) is a scoring system that quantifies disease severity by measuring ocular, bulbar, respiratory and limb strength. The total scores range from 0 to 39, with higher scores indicating greater disease severity.
Change from baseline in the Quantitative Myasthenia Gravis (QMG) score at day 32 | Baseline, Day 32
  The Quantitative Myasthenia Gravis (QMG) is a scoring system that quantifies disease severity by measuring ocular, bulbar, respiratory and limb strength. The total scores range from 0 to 39, with higher scores indicating greater disease severity.
Postinterventional status at day 11 | Day 11
  Postinterventional status is an assessment of whether a participant's MG symptoms/signs have remained unchanged, worsened, improved or reached minimal manifestations or minimal symptom expression.
Postinterventional status at day 18 | Day 18
  Postinterventional status is an assessment of whether a participant's MG symptoms/signs have remained unchanged, worsened, improved or reached minimal manifestations or minimal symptom expression.
Postinterventional status at day 32 | Day 32
  Postinterventional status is an assessment of whether a participants's MG symptoms/signs have remained unchanged, worsened, improved or reached minimal manifestations or minimal symptom expression.
Length of hospital stay | Duration of hospitalization, approximately 7 days
  Length of time between the participant being admitted to discharged. For participants transferred to University of Colorado Hospital, the time of admission/presentation to the outside hospital is counted.
Proportion of participants requiring mechanical ventilation | During hospitalization, approximately 7 days
  Number of participants requiring mechanical ventilation against the total number of participants.
Proportion of participants requiring enteral feeding | During hospitalization, approximately 7 days
  Number of participants requiring enteral feeding (such as an NG tube or PEG tube) against the total number of participants.
Time to freedom from respiratory support | During hospitalization, approximately 7 days
  Length of time between the participant being put on respiratory support (e.g. ventilator, BiPAP) and respiratory support being discontinued.
Change from baseline in Total Immunoglobin G (IgG) at day 32 | Baseline, Day 32
  Immunoglobin G (IgG) total level will be measured via blood collection.
Change from baseline in Acetylcholine Receptor (AchR) antibody titer at day 32 | Baseline, Day 32
  Acetylcholine Receptor (AchR) antibody titer will be measured via blood collection.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ragole, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to NeurologyResearch@cuanschutz.edu. To gain access, data requestors will need to sign a data access agreement.
URL: https://medschool.cuanschutz.edu/neurology/research

REFERENCES:
- [Background] Phillips LH 2nd. The epidemiology of myasthenia gravis. Ann N Y Acad Sci. 2003 Sep;998:407-12. doi: 10.1196/annals.1254.053. PMID 14592908
- [Background] Schneider-Gold C, Hagenacker T, Melzer N, Ruck T. Understanding the burden of refractory myasthenia gravis. Ther Adv Neurol Disord. 2019 Mar 1;12:1756286419832242. doi: 10.1177/1756286419832242. eCollection 2019. PMID 30854027
- [Background] Gilhus NE. Myasthenia Gravis. N Engl J Med. 2016 Dec 29;375(26):2570-2581. doi: 10.1056/NEJMra1602678. No abstract available. PMID 28029925
- [Background] Habib AA, Sacks N, Cool C, Durgapal S, Dennen S, Everson K, Hughes T, Hernandez J, Phillips G. Hospitalizations and Mortality From Myasthenia Gravis: Trends From 2 US National Datasets. Neurology. 2024 Jan 23;102(2):e207863. doi: 10.1212/WNL.0000000000207863. Epub 2023 Dec 18. PMID 38165317
- [Background] Gajdos P, Chevret S, Toyka KV. Intravenous immunoglobulin for myasthenia gravis. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD002277. doi: 10.1002/14651858.CD002277.pub4. PMID 23235588
- [Background] Ipe TS, Davis AR, Raval JS. Therapeutic Plasma Exchange in Myasthenia Gravis: A Systematic Literature Review and Meta-Analysis of Comparative Evidence. Front Neurol. 2021 Aug 31;12:662856. doi: 10.3389/fneur.2021.662856. eCollection 2021. PMID 34531809
- [Background] Gelfand EW. Intravenous immune globulin in autoimmune and inflammatory diseases. N Engl J Med. 2012 Nov 22;367(21):2015-25. doi: 10.1056/NEJMra1009433. No abstract available. PMID 23171098
- [Background] Barth D, Nabavi Nouri M, Ng E, Nwe P, Bril V. Comparison of IVIg and PLEX in patients with myasthenia gravis. Neurology. 2011 Jun 7;76(23):2017-23. doi: 10.1212/WNL.0b013e31821e5505. Epub 2011 May 11. PMID 21562253
- [Background] Guo Y, Tian X, Wang X, Xiao Z. Adverse Effects of Immunoglobulin Therapy. Front Immunol. 2018 Jun 8;9:1299. doi: 10.3389/fimmu.2018.01299. eCollection 2018. PMID 29951056
- [Background] Norda R, Stegmayr BG; Swedish Apheresis Group. Therapeutic apheresis in Sweden: update of epidemiology and adverse events. Transfus Apher Sci. 2003 Oct;29(2):159-66. doi: 10.1016/S1473-0502(03)00121-6. PMID 12941356
- [Background] Kaya E, Keklik M, Sencan M, Yilmaz M, Keskin A, Kiki I, Erkurt MA, Sivgin S, Korkmaz S, Okan V, Dogu MH, Unal A, Cetin M, Altuntas F, Ilhan O. Therapeutic plasma exchange in patients with neurological diseases: multicenter retrospective analysis. Transfus Apher Sci. 2013 Jun;48(3):349-52. doi: 10.1016/j.transci.2013.04.015. Epub 2013 Apr 22. PMID 23619327
- [Background] Francois M, Daubin D, Menouche D, Gaillet A, Provoost J, Trusson R, Arrestier R, Hequet O, Richard JC, Moranne O, Larcher R, Klouche K. Adverse Events and Infectious Complications in the Critically Ill Treated by Plasma Exchange: A Five-Year Multicenter Cohort Study. Crit Care Explor. 2023 Oct 27;5(11):e0988. doi: 10.1097/CCE.0000000000000988. eCollection 2023 Nov. PMID 38304709
- [Background] Bril V, Szczudlik A, Vaitkus A, Rozsa C, Kostera-Pruszczyk A, Hon P, Bednarik J, Tyblova M, Kohler W, Toomsoo T, Nowak RJ, Mozaffar T, Freimer ML, Nicolle MW, Magnus T, Pulley MT, Rivner M, Dimachkie MM, Distad BJ, Pascuzzi RM, Babiar D, Lin J, Querolt Coll M, Griffin R, Mondou E. Randomized Double-Blind Placebo-Controlled Trial of the Corticosteroid-Sparing Effects of Immunoglobulin in Myasthenia Gravis. Neurology. 2023 Feb 14;100(7):e671-e682. doi: 10.1212/WNL.0000000000201501. Epub 2022 Oct 21. PMID 36270895
- [Background] Howard JF Jr, Bril V, Vu T, Karam C, Peric S, Margania T, Murai H, Bilinska M, Shakarishvili R, Smilowski M, Guglietta A, Ulrichts P, Vangeneugden T, Utsugisawa K, Verschuuren J, Mantegazza R; ADAPT Investigator Study Group. Safety, efficacy, and tolerability of efgartigimod in patients with generalised myasthenia gravis (ADAPT): a multicentre, randomised, placebo-controlled, phase 3 trial. Lancet Neurol. 2021 Jul;20(7):526-536. doi: 10.1016/S1474-4422(21)00159-9. PMID 34146511
- [Background] Gwathmey KG, Ding H, Hehir M, Silvestri N. How should newer therapeutic agents be incorporated into the treatment of patients with myasthenia gravis? Muscle Nerve. 2024 Apr;69(4):389-396. doi: 10.1002/mus.28038. Epub 2024 Feb 3. PMID 38308492
- [Background] Ulrichts P, Guglietta A, Dreier T, van Bragt T, Hanssens V, Hofman E, Vankerckhoven B, Verheesen P, Ongenae N, Lykhopiy V, Enriquez FJ, Cho J, Ober RJ, Ward ES, de Haard H, Leupin N. Neonatal Fc receptor antagonist efgartigimod safely and sustainably reduces IgGs in humans. J Clin Invest. 2018 Oct 1;128(10):4372-4386. doi: 10.1172/JCI97911. Epub 2018 Jul 24. PMID 30040076
- [Background] Howard JF Jr, Bril V, Burns TM, Mantegazza R, Bilinska M, Szczudlik A, Beydoun S, Garrido FJRR, Piehl F, Rottoli M, Van Damme P, Vu T, Evoli A, Freimer M, Mozaffar T, Ward ES, Dreier T, Ulrichts P, Verschueren K, Guglietta A, de Haard H, Leupin N, Verschuuren JJGM; Efgartigimod MG Study Group. Randomized phase 2 study of FcRn antagonist efgartigimod in generalized myasthenia gravis. Neurology. 2019 Jun 4;92(23):e2661-e2673. doi: 10.1212/WNL.0000000000007600. Epub 2019 May 22. PMID 31118245
- [Background] Katzberg HD, Barnett C, Merkies IS, Bril V. Minimal clinically important difference in myasthenia gravis: outcomes from a randomized trial. Muscle Nerve. 2014 May;49(5):661-5. doi: 10.1002/mus.23988. Epub 2014 Feb 4. PMID 24810970
- [Background] Guptill JT, Juel VC, Massey JM, Anderson AC, Chopra M, Yi JS, Esfandiari E, Buchanan T, Smith B, Atherfold P, Jones E, Howard JF Jr. Effect of therapeutic plasma exchange on immunoglobulins in myasthenia gravis. Autoimmunity. 2016 Nov;49(7):472-479. doi: 10.1080/08916934.2016.1214823. Epub 2016 Aug 11. PMID 27684107
- [Background] Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology. 1999 Apr 22;52(7):1487-9. doi: 10.1212/wnl.52.7.1487. PMID 10227640
- [Background] Barohn RJ, McIntire D, Herbelin L, Wolfe GI, Nations S, Bryan WW. Reliability testing of the quantitative myasthenia gravis score. Ann N Y Acad Sci. 1998 May 13;841:769-72. doi: 10.1111/j.1749-6632.1998.tb11015.x. No abstract available. PMID 9668327
- [Background] Gajdos P, Tranchant C, Clair B, Bolgert F, Eymard B, Stojkovic T, Attarian S, Chevret S; Myasthenia Gravis Clinical Study Group. Treatment of myasthenia gravis exacerbation with intravenous immunoglobulin: a randomized double-blind clinical trial. Arch Neurol. 2005 Nov;62(11):1689-93. doi: 10.1001/archneur.62.11.1689. PMID 16286541
- [Background] Howard JF Jr, Utsugisawa K, Benatar M, Murai H, Barohn RJ, Illa I, Jacob S, Vissing J, Burns TM, Kissel JT, Muppidi S, Nowak RJ, O'Brien F, Wang JJ, Mantegazza R; REGAIN Study Group. Safety and efficacy of eculizumab in anti-acetylcholine receptor antibody-positive refractory generalised myasthenia gravis (REGAIN): a phase 3, randomised, double-blind, placebo-controlled, multicentre study. Lancet Neurol. 2017 Dec;16(12):976-986. doi: 10.1016/S1474-4422(17)30369-1. Epub 2017 Oct 20. PMID 29066163
- [Background] Vu T, Meisel A, Mantegazza R, Annane D, Katsuno M, Aguzzi R, Enayetallah A, Beasley KN, Rampal N, Howard JF. Terminal Complement Inhibitor Ravulizumab in Generalized Myasthenia Gravis. NEJM Evid. 2022 May;1(5):EVIDoa2100066. doi: 10.1056/EVIDoa2100066. Epub 2022 Apr 26. PMID 38319212
- [Background] Bril V, Druzdz A, Grosskreutz J, Habib AA, Mantegazza R, Sacconi S, Utsugisawa K, Vissing J, Vu T, Boehnlein M, Bozorg A, Gayfieva M, Greve B, Woltering F, Kaminski HJ; MG0003 study team. Safety and efficacy of rozanolixizumab in patients with generalised myasthenia gravis (MycarinG): a randomised, double-blind, placebo-controlled, adaptive phase 3 study. Lancet Neurol. 2023 May;22(5):383-394. doi: 10.1016/S1474-4422(23)00077-7. PMID 37059507
- [Background] Farmakidis C, Pasnoor M, Dimachkie MM, Barohn RJ. Treatment of Myasthenia Gravis. Neurol Clin. 2018 May;36(2):311-337. doi: 10.1016/j.ncl.2018.01.011. PMID 29655452
- [Background] Sharshar T, Porcher R, Demeret S, Tranchant C, Gueguen A, Eymard B, Nadaj-Pakleza A, Spinazzi M, Grimaldi L, Birnbaum S, Friedman D, Clair B; MYACOR Study Group. Comparison of Corticosteroid Tapering Regimens in Myasthenia Gravis: A Randomized Clinical Trial. JAMA Neurol. 2021 Apr 1;78(4):426-433. doi: 10.1001/jamaneurol.2020.5407. PMID 33555314